CLINICAL TRIAL: NCT05555420
Title: Assessment of BMP-2 and ALP Levels Following Laser Therapy as an Adjunct to Scaling and Root Planing for Treatment of Periodontitis- A Randomized Clinical Trial.
Brief Title: BMP-2 and ALP Levels Following Laser Therapy With Scaling and Root Planing in Periodontitis- RCT.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa El Sayed Abbas Ahmed, Dr., Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACU-Dentistry-Perio.1
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Periodontitis, Laser
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SRP only (Active Comparator)
  Interventions: Device: SRP+Laser
- SRP+Laser (Experimental)
  Interventions: Device: SRP+Laser

INTERVENTIONS:
Device: SRP+Laser — Non-surgical periodontal therapy in combination with Laser

SUMMARY:
Patients with periodontitis will be treated by either SRP only or SRP in combination with laser.

Samples from GCF will be collected immediately after treatment and at 3 months follow-up time. Levels of BMP-2 and ALP will be assessed at these time points.

Statistical analysis to compare the results will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis

Exclusion Criteria:

* Uncontrolled medical condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Amount of attachment gain | 3 months
  Described in mm

SECONDARY OUTCOMES:
Level of BMP-2 in GCF | 3 months
  ELISA test
Level of ALP in GCF | 3 months
  Colorimetry